CLINICAL TRIAL: NCT02890836
Title: Blood Pressure, Antihypertensive Treatment and Preeclampsia in Pregnant Wom-en With Pre-existing Diabetes
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Vestgaard, MD, Ph.D student, Rigshospitalet, Denmark
Other Study IDs: H-15019186
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Pregnancy in Diabetics
Keywords: Blood pressure; Hypertension; White coat hypertension; Preeclampsia; Anti-hypertensiva
MeSH Terms: conditions — Pregnancy in Diabetics; Hypertension; White Coat Hypertension; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant women with pre-existing diabetes: Inclusion of 400 women is anticipated.
  Interventions: Drug: Antihypertensiva, mainly Metyldopa
- Healthy pregnant women: Inclusion of 100 women is anticipated

INTERVENTIONS:
Drug: Antihypertensiva, mainly Metyldopa
  Groups: Pregnant women with pre-existing diabetes

SUMMARY:
Aim: First, to investigate the prevalence of a) confirmed hypertension, b) white coat hypertension and c) normal blood pressure in pregnant women with pre-existing diabetes. Second, to explore the prevalence of preeclampsia and preterm delivery in women with pre-existing diabetes with a) confirmed hypertension, b) white coat hypertension and c) normal blood pressure before entering the third trimester of pregnancy. Third, to explore the influence of lifestyle, gestational weight gain and mental well-being on confirmed hypertension and preeclampsia in pregnant women with diabetes.The recruitment period was in 2018 extended to 2020 to perform the following studies: First whether home BP in early pregnancy is superior to office BP to predict preeclampsia. Second to evaluate the prevalence of preeclampsia after initiation of a new treatment strategy including prophylactic aspirin and, in case of insufficiency, vitamin D supplementation.

Design: A prospective multicentre observational study where approximately 400 pregnant women with pre-existing diabetes are offered measurements of office blood pressure (BP) and home BP for three days three times during pregnancy as well as when the routinely measured office BP exceeds 135/85 mmHg. The prevalence of confirmed hypertension (office BP >135/85 mmHg and home BP >130/80 mmHg) and white coat hypertension (office BP >135/85 mmHg but home BP ≤130/80 mmHg) will be determined. Women with confirmed hypertension are offered antihypertensive treatment mainly with methyldopa. In women with a) confirmed hypertension, b) white coat hypertension, and c) normal blood pressure before entering third trimester of pregnancy, the prevalence of preeclampsia and preterm delivery will be evaluated. Possible side effects of antihypertensive treatment including impaired fetal haemodynamics and lower infant birth weight will be recorded. The women will complete food diaries and questionnaires on lifestyle and mental health three times in pregnancy in order to evaluate the influence of these parameters on hypertension and preeclampsia.

DETAILED DESCRIPTION:
Design: Home blood pressure and office blood pressure as predictors of preeclampsia will be evaluated in the total cohort. From February 2018, the routine care includes treatment with prophylactic aspirin in all women with pre-existing diabetes and screening for vitamin D insufficiency, treated with vitamin D depending on the severity of the insufficiency. The prevalence of preeclampsia after initiation of the new treatment strategy will be evaluated. The women included from 2016-2018, where aspirin was only initiated if other risk factors to preeclampsia apart from diabetes were present, will be used for comparison.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for pregnant women with diabetes:

* Women with pre-existing diabetes, older than 18 years and referred to The Center for Pregnant Women with Diabetes, Rigshospitalet, or the Centre for Diabetes and Pregnancy, Odense University Hospital, with a live singleton or twin pregnancy before 20 weeks during the inclusion period.
* Women with diabetes diagnosed in pregnancy before 20 weeks (HbA1c ≥48 mmol/mol) may also be included as having type 2 diabetes.
* Sufficient Danish language skills to read and understand the patient information sheet and to converse.

Inclusion criteria for pregnant healthy women without diabetes:

* Women above 18 years of age, with a live singleton pregnancy, referred to a nuchal translucency scan at 11-14 weeks at The Department of Obstetrics, Rigshospitalet.
* Sufficient Danish language skills to read and understand the patient information sheet and to converse.

Exclusion Criteria:

Exclusion criteria for both study groups:

• Women diagnosed with severe diseases that could possibly bias BP measurements or pregnancy outcome. This is judged by the principal investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohorte of unselected consecutive pregnant women with pre-existing type 1 and type 2 diabetes will be included.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Confirmed hypertension | 2 years
  Office blood pressure >135/85 mmHg measured twice at least 4 hours apart and home blood pressure >130/80 mmHg in pregnancy, or diagnosed hypertension with antihypertensive treatment from before pregnancy
White coat hypertension | 2 years
  Office blood pressure >135/85 mmHg measured twice at least 4 hours apart, but home blood pressure ≤130/80 mmHg
Preeclampsia | 4 years
Early preeclampsia | 4 years
  Preeclampsia occurring before 34 weeks
Preterm birth | 4 years
  Birth before 37 completed weeks
Early preterm delivery (international) | 4 years
  Birth before 32 completed weeks
Early preterm delivery (Danish) | 4 years
  Birth before 34 completed weeks

SECONDARY OUTCOMES:
Gestational hypertension | 4 years
  De novo hypertension appearing after 20 weeks
Chronic hypertension | 4 years
  Hypertension diagnosed prior to pregnancy, or during pregnancy before 20 weeks

OTHER OUTCOMES:
Infant birth weight SD-score | 4 years
Large for gestational age | 4 years
Small for gestational age | 4 years
Ponderal index | 2 years
Gestational weight gain | 4 years
Caesarean section | 4 years
Shoulder dystocia | 4 years
Degree of rupture | 2 years
Duration from induction of labour to delivery | 2 years
Duration of active labour | 2 years
Major congenital malformations | 4 years
  Malformations that include ICD 10 codes: Q00-Q99. In addition, a congenital abnormality that requires medical or surgical treatment, has a serious adverse effect on health and development, or has significant cosmetic impact
Perinatal mortality | 4 years
  Perinatal death includes infant deaths that occur at less than 28 days of age and fetal deaths with a stated or presumed period of gestation of 20 weeks or more
Perinatal morbidity | 4 years
  The occurrence of at least one of the following complications: neonatal hypoglycaemia, neonatal jaundice, transient tachypnea of the newborn or admission to neonatal intensive care unit within the first 28 days of life
Neonatal hypoglycaemia (Danish definition) | 4 years
  Plasma glucose <5 mmol/L, measured within 4 hours of life.
Neonatal hypoglycaemia (common international) | 4 years
  Neonatal hypoglycemia defined as a plasma glucose value < 2.2 mmol/L, measured within 4 hours of life
Jaundice | 4 years
Transient tachypnea of the newborn | 4 years
  A need for Continuous Positive Airway Pressure for more than 60 minutes
Apgar score | 4 years
  A measure of the health of a newborn infant done at 1 and 5 min. The newborn is given points (0, 1, 2) for heart rate, respiratory effort, muscle tone, response to stimulation and skin coloration. A score of 10 points indicates excellent health.
Microalbuminuria | 4 years
  30-300 mg/day albumin or ACR, 30-300 mg/g of creatinine or 3.4-34 mg/mmol of creatinine
Diabetic nephropathy | 4 years
  U-albumin >300 mg/day or albumin to creatinine ratio>300 mg/g of creatinine or >34 mg/mmol of creatinine
Diabetic retinopathy | 4 years
  Presence of any diabetic retinopathy at first examination in pregnancy
Kidney involvement | 4 years
  Diabetic nephropathy or microalbuminuria
Pulsatility index (PI) of the middle cerebral artery (MCA) measured with Doppler flow measurements | 2 years
Pulsatility index (PI) of the umbilical artery (UA) measured with Doppler flow | 2 years
Ratio of the pulsatility index (PI) of the middle cerebral artery and the umbilical artery | 2 years
Body mass index (BMI) | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Pregnant Women with Diabetes, Copenhagen, Kbh Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Do NC, Vestgaard M, Asbjornsdottir B, Andersen LLT, Jensen DM, Ringholm L, Damm P, Mathiesen ER. Home Blood Pressure for the Prediction of Preeclampsia in Women With Preexisting Diabetes. J Clin Endocrinol Metab. 2022 Aug 18;107(9):e3670-e3678. doi: 10.1210/clinem/dgac392. PMID 35766641
- [Derived] Asbjornsdottir B, Vestgaard M, Do NC, Ringholm L, Andersen LLT, Jensen DM, Damm P, Mathiesen ER. Prevalence of anxiety and depression symptoms in pregnant women with type 2 diabetes and the impact on glycaemic control. Diabet Med. 2021 Mar;38(3):e14506. doi: 10.1111/dme.14506. Epub 2021 Jan 8. PMID 33368557
- [Derived] Do NC, Vestgaard M, Asbjornsdottir B, Nichum VL, Ringholm L, Andersen LLT, Jensen DM, Damm P, Mathiesen ER. Physical activity, sedentary behavior and development of preeclampsia in women with preexisting diabetes. Acta Diabetol. 2020 May;57(5):559-567. doi: 10.1007/s00592-019-01459-7. Epub 2019 Nov 28. PMID 31781957
- [Derived] Vestgaard M, Asbjornsdottir B, Ringholm L, Andersen LLT, Jensen DM, Damm P, Mathiesen ER. White coat hypertension in early pregnancy in women with pre-existing diabetes: prevalence and pregnancy outcomes. Diabetologia. 2019 Dec;62(12):2188-2199. doi: 10.1007/s00125-019-05002-9. Epub 2019 Oct 18. PMID 31628489